CLINICAL TRIAL: NCT07362420
Title: Effects of Myofascial Chain-Based Specific Exercise and Myofascial Trigger Point Therapy in People With Non-Specific Low Back Pain
Brief Title: Comparing Myofascial Exercise and Trigger Point Therapy for Non-Specific Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Wendy Tzyy-Jiuan Wang, Professor, Department of Physical Therapy, National Yang Ming Chiao Tung University, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU114206AE
Record Dates: First submitted 2026-01-07; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Non-specific Low Back Pain
Keywords: Non-specific Low Back Pain; Low Back Pain; Myofascial Trigger Points; Myofascial Chain; Exercise Therapy; Manual Therapy; Physical Therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Myofascial Trigger Point Manual Compression Group (Experimental): Participants in this group receive myofascial trigger point manual compression only. A licensed physical therapist applies sustained manual pressure to identified myofascial trigger points using standardized, noninvasive procedures.
  Interventions: Other: Myofascial Trigger Point Manual Compression
- Myofascial Chain-Based Specific Exercise Group (Experimental): Participants in this group receive a myofascial chain-based specific exercise program only. The supervised exercise program is delivered by a physical therapist and focuses on movement control and muscle function within targeted myofascial chains.
  Interventions: Other: Myofascial Chain-Based Specific Exercise
- Combined Manual Compression and Exercise Group (Experimental): Participants in this group receive a combined intervention consisting of myofascial trigger point manual compression followed by a myofascial chain-based specific exercise program within the same treatment session.
  Interventions: Other: Myofascial Trigger Point Manual Compression; Other: Myofascial Chain-Based Specific Exercise

INTERVENTIONS:
Other: Myofascial Trigger Point Manual Compression — This intervention consists of noninvasive hands-on manual pressure applied by a licensed physical therapist to identified myofascial trigger points associated with nonspecific low back pain. Treatment sessions are provided twice per week over a four-week period. Manual compression is applied using standardized clinical procedures at an intensity tolerated by the participant. The selection of trigger points follows predefined criteria to ensure consistency across treatment sessions.
  This intervention is noninvasive and does not involve the use of any drugs or medical devices.
  Arms: Combined Manual Compression and Exercise Group; Myofascial Trigger Point Manual Compression Group
Other: Myofascial Chain-Based Specific Exercise — This intervention is a supervised, noninvasive exercise program delivered by a licensed physical therapist. Participants attend exercise sessions twice per week for four weeks. The program focuses on movement control and muscle function within targeted myofascial chains and is tailored based on functional muscle performance. Exercise selection and progression follow standardized clinical criteria to promote safe and consistent implementation.
  This intervention is noninvasive and does not involve the use of any drugs or medical devices.
  Arms: Combined Manual Compression and Exercise Group; Myofascial Chain-Based Specific Exercise Group

SUMMARY:
The goal of this clinical trial is to learn if two common physical therapy approaches, used alone or together, can help reduce pain and improve daily function in adults with nonspecific low back pain. Nonspecific low back pain means low back pain without a clear medical cause.

The main questions this study aims to answer are:

1. Does hands-on pressure to painful muscle spots (called myofascial trigger point therapy) help lower low back pain?
2. Does a guided exercise program that focuses on how muscles work together help lower low back pain?
3. Does combining hands-on therapy with exercise work better than using either approach alone?

Researchers will compare three groups to see which approach leads to greater improvement. One group will receive hands-on trigger point therapy, one group will do a specific exercise program, and one group will receive both treatments.

Participants will:

* Be assigned to one of the three treatment groups by chance
* Receive treatment twice a week for four weeks
* Complete simple assessments before treatment starts, after the first treatment session, and after the final session

The results of this study may help physical therapists choose better noninvasive treatment options for people with nonspecific low back pain.

DETAILED DESCRIPTION:
Non-specific low back pain is common, recurrent, and associated with substantial disability and health care use. In people with persistent symptoms, myofascial trigger points (MTrPs) are frequently identified and may contribute to heightened local pain sensitivity, restricted movement, and altered muscle recruitment patterns. In parallel, impaired kinetic-chain function and deficits in neuromuscular control are widely considered clinically relevant in nonspecific low back pain. From a myofascial perspective, regional symptoms may be influenced by force transmission and coordination across interconnected tissues and muscles within myofascial chains, particularly those spanning the trunk and lower extremity.

This trial is grounded in a combined framework that integrates (1) a local, noninvasive manual approach targeting MTrP-related pain sensitivity and mechanical irritability and (2) a function-oriented, myofascial chain-based exercise approach designed to address movement dysfunction and chain-level performance. The exercise program applies a functional classification model distinguishing stabilizer and mobilizer muscle roles. Stabilizer dysfunction is addressed through low-load inner-range holding strategies aimed at improving segmental control and endurance, whereas mobilizer dysfunction is addressed through sustained stretching strategies aimed at improving available range and reducing compensatory movement patterns. The central hypothesis is that combining these two approaches may provide complementary benefits by first reducing local pain sensitivity and then consolidating gains through task-relevant neuromuscular retraining and chain-based loading.

This study is an assessor-blinded, three-arm randomized controlled trial. Adults with nonspecific low back pain will be randomized to receive either (1) MTrP manual compression, (2) myofascial chain-based specific exercise, or (3) a combined intervention. Interventions will be delivered by trained physical therapists using standardized, protocol-driven procedures, twice weekly over four weeks. The protocol includes decision rules intended to standardize session content while allowing limited adjustment to individual presentation (e.g., selection of the most clinically relevant trigger point per target muscle and tailoring of exercise progression based on movement quality and compensations).

To evaluate both immediate and overall intervention effects, assessments will be conducted at three time points: prior to the first treatment session (baseline), immediately after the first session (immediate response), and after completion of the final treatment session (post-intervention). The outcomes are selected to reflect pain sensitivity, function and disability, and mechanistic/functional domains relevant to the study framework (e.g., chain-level performance, neuromuscular function, and lumbar movement capacity). Home program adherence will be monitored with participant logs for exercise-containing groups, supporting interpretation of treatment response in relation to dosage and compliance.

Treatment fidelity will be supported through therapist training, use of standardized procedures, and documentation of session content and dosage. Safety monitoring will be conducted throughout the intervention period. Because all interventions are noninvasive and commonly used in physical therapy practice, major adverse events are not expected; however, any discomfort, symptom exacerbation, or other adverse responses will be recorded and managed according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years
* Nonspecific low back pain lasting longer than 6 weeks
* Average low back pain intensity of 3 or higher on a 0-10 Numeric Pain Rating Scale
* Presence of at least 6 myofascial trigger points identified across bilateral target muscles
* Presence of muscle function impairments in at least 6 muscle groups based on functional muscle testing
* Able to understand study procedures and participate in an exercise-based intervention
* Willing and able to attend treatment sessions and complete study assessments

Exclusion Criteria:

* Currently pregnant
* Diagnosed spondylolisthesis or vertebral compression fracture
* Known malignancy or history of cancer affecting the spine
* Previous lumbar spine surgery
* Known neurological, infectious, or systemic disease that may affect pain or movement
* Any other medical condition that, in the opinion of the investigators, would interfere with safe participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline (before the first treatment session), immediately after the first treatment session, and after the final treatment session (4 weeks)
  Pain intensity is assessed using the Numeric Pain Rating Scale (NPRS). Participants rate their current low back pain on an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable). Lower scores indicate less pain.

SECONDARY OUTCOMES:
Functional performance | Baseline (before the first treatment session) and after the final treatment session (4 weeks)
  Functional performance is assessed using the Patient-Specific Functional Scale (PSFS). Participants identify activities limited by low back pain and rate their ability to perform each activity on a scale from 0 (unable to perform) to 10 (able to perform without difficulty). Higher scores indicate better function.
Low Back Pain-Related Disability | Baseline (before the first treatment session) and after the final treatment session (4 weeks)
  Disability related to low back pain is assessed using the Oswestry Disability Index (ODI). The ODI measures the impact of low back pain on daily activities, with higher scores indicating greater disability.
  The Oswestry Disability Index (ODI) was used in this study to assess the level of disability in individuals with low back pain. The ODI consists of ten items designed to quantify the impact of low back pain on activities of daily living. Each item includes six statements, scored from 0 to 5, with 0 indicating no pain, no difficulty, and no functional limitation, and 5 indicating severe pain or disability that prevents the performance of the activity. The total score is calculated as a percentage, with 0% representing no disability and **100% representing the highest level of disability.
Myofascial Chain Extensibility | Baseline (before the first treatment session) and after the final treatment session (4 weeks)
  Myofascial chain extensibility is assessed using standardized extensibility tests targeting three myofascial chains: the Superficial Back Line, Front Functional Line, and Back Functional Line.
  Superficial Back Line extensibility is assessed using a standing forward-bending test, with the distance between the fingertips and the ground measured in centimeters.
  Front Functional Line extensibility is assessed using a lunge-based trunk rotation test, with trunk rotation angle measured in degrees.
  Back Functional Line extensibility is assessed using a kneeling side-bending posture, with thoracolumbar side-bending angle measured in degrees using a goniometer.
Myofascial Chain Endurance | Baseline (before the first treatment session) and after the final treatment session (4 weeks)
  Myofascial chain endurance is assessed using standardized endurance tests targeting three myofascial chains: the Superficial Back Line, Front Functional Line, and Back Functional Line.
  Superficial Back Line endurance is assessed using a modified Sorensen test, in which participants maintain a horizontal trunk position until voluntary fatigue occurs, without the presence of pain or compensatory movement.
  Front Functional Line endurance is assessed using a supine abdominal curl-up endurance test with lower-limb adduction, with time recorded until voluntary fatigue occurs, without pain or compensatory movement.
  Back Functional Line endurance is assessed using a modified quadruped endurance test, with participants maintaining simultaneous upper- and lower-limb elevation until voluntary fatigue occurs, without pain or compensatory movement.
Muscle Function | Baseline (before the first treatment session) and after the final treatment session (4 weeks)
  Muscle function is evaluated using standardized clinical tests to assess stabilizer and mobilizer muscle performance. Test results indicate the ability to maintain controlled isometric contraction or complete functional movement without compensation.
  Stabiliser muscle testing was performed for the psoas major and gluteus maximus, while mobiliser muscle testing was conducted for the hamstrings, quadratus lumborum, latissimus dorsi, iliocostalis lumborum, adductor longus, rectus abdominis, pectoralis major, and gastrocnemius.
  For stabiliser muscles, the assessment evaluated whether the muscle could maintain a stable isometric contraction within its intrinsic functional range for 15 seconds, repeated twice, while monitoring for the presence of compensatory movements.
  For mobiliser muscles, the assessment evaluated whether the muscle could be brought through its maximal functional range of motion, with observation for any compensatory movements.
Lumbar Active Range of Motion | Baseline (before the first treatment session), immediately after the first treatment session, and after the final treatment session (4 weeks)
  Lumbar active range of motion is measured in flexion, extension, side bending, and rotation using a back range-of-motion measurement (BROM II) device. Greater values indicate increased lumbar mobility.
Central Sensitization | Baseline (before the first treatment session) and after the final treatment session (4 weeks)
  Central sensitization is assessed using the Central Sensitization Inventory (CSI), a self-report questionnaire measuring symptoms related to pain sensitization. Higher scores indicate greater central sensitization.
  Participants answer a series of questions about symptoms related to central sensitization, rating each item from 0 (never) to 4 (always). A score of more than 40 indicates the presence of central sensitisation.
Pressure Pain Threshold | Baseline (before the first treatment session), immediately after the first treatment session, and after the final treatment session (4 weeks)
  Pressure pain threshold is measured using a handheld algometer applied to selected myofascial trigger points. Higher values indicate lower pain sensitivity.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share individual participant data. This decision may be re-evaluated upon study completion or at the time of publication.